CLINICAL TRIAL: NCT02576418
Title: Evaluation of the PartoSure Time to Delivery (TTD) Test to Predict Spontaneous Preterm Delivery in Pregnancies After Assisted Reproductive Technology (ART)
Brief Title: PartoSure to Predict Spontaneous Preterm Delivery in Pregnancies After Assisted Reproductive Technology (ART)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vietnam National University (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_08_2015
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Infertility
Keywords: Partosure TTD test; CL; ART; SN; SP; PPV; NPV
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Partosure TTD Test (Experimental): PartoSure TTD test will be performed on all patients and the test-to-spontaneous-delivery interval will be calculated.
  Interventions: Other: Partosure TTD test

INTERVENTIONS:
Other: Partosure TTD test — PartoSure TTD test and CL will be performed on all patients and the test-to-spontaneous-delivery interval will be calculated.

SUMMARY:
To calculate sensitivity (SN), specificity (SP), positive predictive value (PPV) and negative predictive value (NPV) of PartoSure TTD test in predicting delivery within 7 or 14 days from testing and to compare it with cervical length (CL) measurement by transvaginal ultrasound (15 mm cut-off)

DETAILED DESCRIPTION:
* This trial is a prospective observational study.
* Pregnancies after ART between 20 0/7 and 36 6/7 weeks with symptoms of preterm labor, clinically intact membranes, cervical dilatation of ≤ 2 cm will be invited to participate to the study. Signed consent form is required to be able to participate to the study.
* PartoSure and CL will be performed on all patients and the test-to-spontaneous-delivery interval will be calculated.
* Trial Population:Pregnancies after ART between 20 0/7 and 36 6/7 weeks with symptoms of preterm labor are hospitalized at My Duc hospital from October 2015 to April 2016. The sample size for this trial of 100 subjects.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment into this trial, each female subject must fulfill all of the following criteria at the start of enrollment:

* Pregnancies after assisted reproductive technology include singleton and twins
* Between 20 0/7 and 36 6/7 weeks with symptoms of preterm labor including uterine contractions, intermittent lower abdominal pain and pelvic pressure.
* Clinically intact membranes.
* Cervical dilatation of ≤ 2 cm
* Agree to participate in the study, and to disclose any medical events to the investigator
* Have given written informed consent

Exclusion Criteria:

To be eligible for enrollment in this study each subject must not meet any of the following criteria:

* Vaginal bleeding
* Overt rupture of the fetal membranes as indicated by visualized leakage of fluid from the cervix
* Placenta previa
* Cervical cerclage in place
* Received tocolytic medications for treatment of threatened preterm delivery prior to collection of the cervicovaginal specimens or CL measurement.
* Digital exam prior to specimen collection.
* A symptom not associated with idiopathic threatened preterm delivery (e.g trauma)
* Enrollment in a tocolytic study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The accuracy of c(SN, SP, PPV, NPV) in predicting delivery within 7 or 14 days from testing | 7 or 14 days from testing
  SN, SP, PPV and NPV superiority of PartoSure TTD test compared to CL measurement via transvaginal ultrasound (15 mm cutoff) for the presentation-to-spontaneous-delivery time intervals of ≤ 7 days or 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, Doctor, Study Director — Research Center for Genetics and Reproductive Health
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ward 13. Tan Binh District, Vietnam